CLINICAL TRIAL: NCT00263627
Title: A Multicentre Randomised Placebo-controlled Double-blind Clinical Trial for Evaluation of Safety and Efficacy of Specific Immunotherapy With an Aluminium Hydroxide-adsorbed Allergoid Preparation of Birch Pollen Allergens
Brief Title: Safety and Efficacy of Specific Immunotherapy With an Aluminium Hydroxide-adsorbed Allergoid Preparation of Birch Pollen Allergens
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Al0204AV; 2005-000025-35 (EudraCT Number)
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2013-11

CONDITIONS: Pollen Allergy
Keywords: specific immunotherapy; birch pollen allergy; Allergovit
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Sterile aluminium hydroxide suspension for subcutaneous injection were applied in the upper arm. Vials with strength A contained 0.0125 mg/mL and with strength B 0.125 mg/mL histamine-dihydrochloride and strength 0 was produced by dilution of strength A. The vials containing the placebo solution were identical in their outer appearance with the active study preparation of the birch pollen allergoids.
  Interventions: Other: Placebo
- Specific Immunotherapy (Experimental): Subcutaneous injections with birch pollen allergoid were applied in the upper arm. Vials with three different concentrations were used: Strength A (1000 TU/mL), strength B (10 000 TU/mL) and strength 0 (100 TU/mL) by dilution of strength A.
  Interventions: Biological: Birch pollen allergoid

INTERVENTIONS:
Biological: Birch pollen allergoid — Subcutaneous injections were applied in the upper arm. Vials with three different concentrations were used: Strength A (1000 TU/mL), strength B (10 000 TU/mL) and strength 0 (100 TU/mL) by dilution of strength A.
  Other Names: specific immunotherapy
  Arms: Specific Immunotherapy
Other: Placebo — Sterile aluminium hydroxide suspension for subcutaneous injection were applied in the upper arm. Vials with strength A contained 0.0125 mg/mL and with strength B 0.125 mg/mL histamine-dihydrochloride and strength 0 was produced by dilution of strength A. The vials containing the placebo solution were identical in their outer appearance with the active study preparation of the birch pollen allergoids.
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to show safety and efficacy of the allergoid preparation of birch pollen allergens in the treatment of birch allergic patients in a representative number of patients.

DETAILED DESCRIPTION:
Type I allergy is an immune-disorder which stems from the formation of IgE antibodies against proteins and glycoproteins from plants, insects, animals and fungi, most of which for healthy subjects are considered to be harmless. However, in allergic patients the cross-linking of specific IgE-antibodies on effector cells by allergens activates an immunological cascade leading to the symptoms of Type I allergy including rhinitis, conjunctivitis, asthma, and anaphylactic shock. Pollens from wind-pollinated plants including trees, grasses and weeds, are amongst the most frequent and potent elicitors of Type I allergy. It is not possible to avoid exposure to these pollens and therefore the symptoms that patients inevitably suffer must be treated with either symptomatic medication or allergen specific immunotherapy.

The Betulaceae family includes the genera Alnus (alder), Betula (birch) and Corylus (hazel). Trees belonging to these genera are widespread in middle and northern Europe and, in combination with the fact that they shed large quantities of wind-borne pollen, leads to their allergenic significance. The prevalence of sensitisation to birch pollen has been studied, and in the case of a middle European (Viennese) population, for example, it has been demonstrated that approximately 40 % of patients with allergic rhinitis are sensitised. Although the pollen season for any one genera seldom lasts for more than a few weeks, the well-documented cross-reactivity between the different Betulaceae and other tree pollens of the Fagales order contributes to a protracted season of symptoms for many allergic patients.

Allergoids are prepared by chemical modification of partially purified native aqueous aller-gen extracts. Native allergen extracts are depleted of components with a molecular mass of less than 5000 Dalton by diafiltration prior to chemical modification with aldehydes. The modification causes a substantial reduction in the allergenicity of the extract as can be judged by skin prick testing, provocation testing, histamine release from sensitised leukocytes and measurement of IgE-binding activity by RAST-inhibition. However, immunogenic activity and T-cell reactivity are retained. These properties enable allergoids to be used as a basis for allergen specific immunotherapy with a reduced risk of inducing IgE-mediated side-reactions and the possibility of administering larger doses of immunogen over a shorter time course than with native allergens.

ELIGIBILITY:
Inclusion Criteria:

* Rhinitis
* Rhinoconjunctivitis
* Positive skin prick test to birch pollen
* Positive radioallergosorbent test (RAST) to birch pollen
* Positive provocation test result to birch pollen

Exclusion Criteria:

* Serious chronic diseases
* Other perennial allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 253 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Symptom Medication Score (SMS) | over a period of eight to twelve weeks during the two pollen seasons in
  The primary endpoint was the area under the curve (AUC) of the daily sum of the Symptom Medication Score (SMS) after two years of double-blind treatment. Each patient recorded the information used for deriving the SMS over a period of eight to twelve weeks during the two double-blind pollen seasons in 2006 and 2007.

SECONDARY OUTCOMES:
Adverse events (AEs) | Entrire study period.
  Safety: (all five years of treatment) occurrence of adverse events (AEs).

OTHER OUTCOMES:
Well days | Entire diary period
  Number of "well days" (Symptom Score ≤ 4, Medication Score = 0)

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Narkus, M.D., Principal Investigator
Locations (1):
- Allergopharma Joachim Ganzer KG, Reinbek, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2005-000025-35/DE